CLINICAL TRIAL: NCT00347698
Title: Intravitreal Bevacizumab vs Panretinal Photocoagulation for the Treatment of Proliferative Diabetic Retinopathy: A One-year Prospective, Contralateral Eye Study
Brief Title: Intravitreal Bevacizumab vs Photocoagulation for Proliferative Diabetic Retinopathy
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Undefined.
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APEC-007
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; bevacizumab; photocoagulation
MeSH Terms: conditions — Diabetic Retinopathy

INTERVENTIONS:
Drug: intravitreal injection of bevacizumab
Procedure: panretinal photocoagulation

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of 2.5 mg of intravitreal bevacizumab in one eye, versus panretinal photocoagulation in the contralateral eye, for the treatment of patients with untreated symmetric proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
The current gold standard for the treatment of proliferative diabetic retinopathy is panretinal photocoagulation. However, it is a treatment that results in significant discomfort to the patient, causes reduction of visual acuity and visual field impairment. Intravitreal bevacizumab is a novel treatment that reduces intraocular VEGF concentration and therefore inhibits neovascular proliferation, without causing significant disconfort to the patient, nor affecting visual acuity or visual fields (although with other risks associated with intravitreal injection). Making a comparison between both treatments in different patients is difficult because there are other variables that influence the progression of the disease (such as glycemic control or renal insufficiency). Therefore this study is designed using both treatments in the same patient: intravitreal bevacizumab in one eye, compared to panretinal photocoagulation in the contralateral eye, and evaluating visual acuity, visual fields, fluorescein angiography, optic coherence tomography of the macula, and patient discomfort, in a one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* symmetric proliferative diabetic retinopathy without high risk characteristics
* age 18 years or older
* patient consent

Exclusion Criteria:

* heart attack or cerebrovascular attack
* only eye
* retinal detachment
* vitreous haemorrhage
* previous treatment for diabetic retinopathy
* media opacities that preclude visualization of the fundus
* pregnancy
* inability to understands the implications of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2006-03 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity at six months and one year
Macular thickness measured by OCT at six months and one year
Median deviation in visual fields at one year
Score on a patient satisfaction scale at six months and one year

SECONDARY OUTCOMES:
Complications associated to each treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo García-Aguirre, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación para Evitar la Ceguera en México, Mexico City, D. F, Mexico

REFERENCES:
- [Background] Treatment techniques and clinical guidelines for photocoagulation of diabetic macular edema. Early Treatment Diabetic Retinopathy Study Report Number 2. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1987 Jul;94(7):761-74. doi: 10.1016/s0161-6420(87)33527-4. PMID 3658348
- [Background] Frank RN. Visual fields and electroretinography following extensive photocoagulation. Arch Ophthalmol. 1975 Aug;93(8):591-8. doi: 10.1001/archopht.1975.01010020575004. PMID 1171677
- [Background] Salti H. Visual dysfunction after panretinal photocoagulation in patients with severe diabetic retinopathy and good vision. Am J Ophthalmol. 2006 Feb;141(2):422; author reply 422-3. doi: 10.1016/j.ajo.2005.10.040. No abstract available. PMID 16458724
- [Background] Witmer AN, Vrensen GF, Van Noorden CJ, Schlingemann RO. Vascular endothelial growth factors and angiogenesis in eye disease. Prog Retin Eye Res. 2003 Jan;22(1):1-29. doi: 10.1016/s1350-9462(02)00043-5. PMID 12597922
- [Background] Presta LG, Chen H, O'Connor SJ, Chisholm V, Meng YG, Krummen L, Winkler M, Ferrara N. Humanization of an anti-vascular endothelial growth factor monoclonal antibody for the therapy of solid tumors and other disorders. Cancer Res. 1997 Oct 15;57(20):4593-9. PMID 9377574
- [Background] Spaide RF, Fisher YL. Intravitreal bevacizumab (Avastin) treatment of proliferative diabetic retinopathy complicated by vitreous hemorrhage. Retina. 2006 Mar;26(3):275-8. doi: 10.1097/00006982-200603000-00004. PMID 16508426
- [Background] Avery RL. Regression of retinal and iris neovascularization after intravitreal bevacizumab (Avastin) treatment. Retina. 2006 Mar;26(3):352-4. doi: 10.1097/00006982-200603000-00016. No abstract available. PMID 16508438
- [Background] Iturralde D, Spaide RF, Meyerle CB, Klancnik JM, Yannuzzi LA, Fisher YL, Sorenson J, Slakter JS, Freund KB, Cooney M, Fine HF. Intravitreal bevacizumab (Avastin) treatment of macular edema in central retinal vein occlusion: a short-term study. Retina. 2006 Mar;26(3):279-84. doi: 10.1097/00006982-200603000-00005. PMID 16508427
- [Background] Rosenfeld PJ, Moshfeghi AA, Puliafito CA. Optical coherence tomography findings after an intravitreal injection of bevacizumab (avastin) for neovascular age-related macular degeneration. Ophthalmic Surg Lasers Imaging. 2005 Jul-Aug;36(4):331-5. PMID 16156152
- [Background] Rosenfeld PJ, Fung AE, Puliafito CA. Optical coherence tomography findings after an intravitreal injection of bevacizumab (avastin) for macular edema from central retinal vein occlusion. Ophthalmic Surg Lasers Imaging. 2005 Jul-Aug;36(4):336-9. PMID 16156153